CLINICAL TRIAL: NCT02729402
Title: Evaluation of the Impact of Cochlear Implants on Cognition in Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Richard Gurgel, MD, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 83983
Record Dates: First submitted 2015-11-04; First posted 2016-04-06 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Dementia; Hearing Loss; Presbycusis
Keywords: Adults
MeSH Terms: conditions — Dementia; Hearing Loss; Presbycusis | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Older Cochlear Implant Subjects (Experimental): We will assign the study participants to a diagnostic intervention (cognitive testing) before and after their cochlear implant.
  Interventions: Other: Cognitive Testing

INTERVENTIONS:
Other: Cognitive Testing — We will use a battery of neurocognitive tests to assess cognitive function before and after surgery

SUMMARY:
The subjects will be age 65 years and older, with no upper limit of age range with hearing loss that are candidates for standard-of-care cochlear implant.

Cognitive tests will be administered preoperative, and postoperative at 6 and 12 month intervals.

DETAILED DESCRIPTION:
Patients >65 year old who are cochlear implant candidates will be recruited for study participation. Candidacy criteria will be based on current FDA guidelines for cochlear implantation. After pre-operative cognitive testing, subjects will undergo cochlear implantation using standard operative techniques. Patient will have routine post-operative care and will follow up with audiology per standard post-activation routine - 1 week after activation, then monthly until a stable program is achieved. Hearing will be measured with standard audiometry to check for residual acoustic hearing, hearing in noise tests (HINT), aided thresholds, and consonant-nucleus-consonant (CNC) words at activation, 6 and 12 months post-operatively, and as often as needed in the interim to determine function.

Pre-operative and 6 and 12 month post-operative cognitive testing will be performed using a battery of tests that will differentiate verbal/auditory and non-verbal cognitive abilities.

Written informed consent will be sought from all individuals who will participate in the proposed project. Consent will be obtained by the principal investigator or key study personnel such as the research coordinator. When a potential participant has been identified, she/he will be visited in person. The participant will be given an overview of the study as well as written material that further explains the study and the responsibilities of the participant. Since some of our participants may have cognitive impairment, we will also make a determination about capacity to provide informed consent. Following presentation of the informed consent document, participants will be asked questions about the study (i.e. purpose, procedures, risks, and benefits). If these questions are adequately answered, then the participant will be judged to have capacity to provide informed consent. However, if these questions are not adequately answered, the participants will not be judged to have this capacity. In these latter cases, assent will be obtained from the participant and informed consent will be obtained from the participant's legally authorized representative (spouse, adult child

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be age 65 years and older, with no upper limit of age range with hearing loss that are candidates for a cochlear implant.

Exclusion Criteria:

* Those patients who are not able to undergo cochlear implantation surgery due to medical co-morbidities would not be eligible for the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-11; Primary Completion 2025-03 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
What is impact on cognition of a cochlear implant in older adults | 4 years
  We will measure cognitive function by administering the mini-mental status exam (MMSE).
What is impact on cognition of a cochlear implant in older adults | 4 years
  We will measure cognitive function by administering the D2 test.
What is impact on cognition of a cochlear implant in older adults | 4 years
  We will measure cognitive function by administering the Hopkins Verbal Learning Test (HVLT) test.
What is impact on cognition of a cochlear implant in older adults | 4 years
  We will measure cognitive function by administering the Digit Span vs. Spatial Span test.
What is impact on cognition of a cochlear implant in older adults | 4 years
  We will measure cognitive function by administering the Hayling Sentence Completion test.
What is impact on cognition of a cochlear implant in older adults | 4 years
  We will measure cognitive function by administering the Stroop Color Word test.
What is impact on cognition of a cochlear implant in older adults | 4 years
  We will measure cognitive function by administering the Brief Visuospatial Memory test.
What is impact on cognition of a cochlear implant in older adults | 4 years
  We will measure cognitive function by administering the Trails A/B test.

SECONDARY OUTCOMES:
What is the psychosocial impact of cochlear implants on older adults | 4 years
  We will measure psychosocial well being (i.e. depression and social interaction) by using the Geriatric depression scale on psychosocial status will be administered

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gurgel, MD, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: No